CLINICAL TRIAL: NCT02822976
Title: The Association Between Glycosylated Hemoglobin A1c (HbA1c) and Outcomes in the Critically Ill
Brief Title: HbA1c and Outcomes in the Critically Ill
Status: Completed | Type: Observational
Sponsor: Roupen Hatzakorzian, MD (Other)
Responsible Party: Sponsor-Investigator, Roupen Hatzakorzian, MD, Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Other Study IDs: 10-276-BMA
Record Dates: First submitted 2015-06-22; First posted 2016-07-06 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Critically Ill Patient HbA1c<6.5: Patients admitted to an intensive care unit with a HbA1c <6.5.
- Critically Ill Patient HbA1c≥6.5: Patients admitted to an intensive care unit with a HbA1c ≥6.5.

SUMMARY:
Background: Glycated hemoglobin A1c (HbA1c) has been linked to poor outcomes in the cardiac surgery, septic and critically ill patient population. It is a promising test to understand the complex relationship between glycemia, diabetes and outcomes in patients admitted to the intensive care unit.

Hypothesis: An elevated HbA1c value on admission to an intensive care unit (ICU) is associated with poor outcomes.

DETAILED DESCRIPTION:
Objectives: The primary objective of this study is to determine hospital mortality of all newcomers admitted to the ICU, and to compare it between patients with HbA1c <6.5% and ≥6.5%. Other outcomes that will be measured include ICU and one year mortality, ICU and hospital length of stay (LOS), days on mechanical ventilation, serious infection during hospitalization and renal failure requiring dialysis during hospitalization and at 6 months. The investigators will also determine the prevalence of pre-diabetes (HbA1c 6.0-6.4%) and diabetes (≥6.5%) in the critically ill population based on HbA1c levels and monitor glucose control and insulin requirements during the first three days of ICU admission.

Methods: This project is a prospective observational study at the McGill University Health Center adult medical and surgical ICUs. HbA1c is measured at the admission to the ICU. The data are being collected prospectively using Microsoft access data entry. The following parameters will be recorded on admission: admitting diagnosis, sex, age, height, weight, body mass index (BMI), Acute Physiology and Chronic Health Evaluation (APACHE) II score, previous diagnosis of DM, whole blood HbA1c level, blood and plasma glucose levels. With power 80%, type I error 5% and with an expected 25% mortality difference between patients with HbA1c≥6.5 and <6.5, the required sample size is 1800 patients. The data will be presented as mean ± SD unless otherwise specified and statistical significance will be set as P < 0.05. All p-values presented will be 2-tailed.

Significance: The investigators want to demonstrate that HbA1c ≥6.5 on admission to an intensive care unit is associated with increased 6 month mortality and worse outcomes. The investigators will also determine the prevalence of pre-diabetes and diabetes in the critically ill based on HbA1c.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to an intensive care unit within 48 hours

Exclusion Criteria:

* Patients with known hemoglobinopathy(ies)
* Patients that have received ≥2 units of packed red blood cells 48 hours prior to HbA1c sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All newcomers to the the McGill University Health Center adult medical and surgical ICUs.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2011-09; Primary Completion 2015-07 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Hospital mortality | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks

SECONDARY OUTCOMES:
ICU mortality | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
One year mortality | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
ICU and Hospital Length of Stay | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
Days on Mechanical Ventilation | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
Serious infections | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
Renal failure requiring dialysis | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks

OTHER OUTCOMES:
Prevalence of pre-diabetes and diabetes in the critically ill | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roupen Hatzakorzian, MD, MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre: Royal Victoria Hospital and Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes